CLINICAL TRIAL: NCT03772652
Title: Long-term Surgical Therapeutic Outcomes of Peri-Implantitis
Status: Terminated | Type: Observational
Why Stopped: COVID-19 pandemic
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Hom-Lay Wang, DDS, MSD, Ph D, Collegiate Professor of Periodontics and Professor of Dentistry, University of Michigan
Other Study IDs: HUM00148346
Record Dates: First submitted 2018-12-05; First posted 2018-12-11 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2021-12

CONDITIONS: Peri-Implantitis
MeSH Terms: conditions — Peri-Implantitis | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Peri-implantitis: Subjects who were diagnosed with peri-implantitis and received treatment at least five years ago at the Graduate Periodontics Clinic at University of Michigan with sufficient baseline data. Soft tissue measurements (observation) of the implant will be completed.
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — Soft tissue implant measurements

SUMMARY:
This study focuses on evaluating the success of different treatment methods for peri-implantitis (gum disease around implants) and to understand the factors that might affect the success of the treatment provided.

DETAILED DESCRIPTION:
Qualifying patients will be asked to participate in clinical measurements to compare the long-term success of their treatments.

The aims of the current study are to 1) assess the long-term outcome of the surgical treatment of peri-implantitis and to 2) evaluate the success of the different treatment modalities of peri-implantitis.

ELIGIBILITY:
Inclusion Criteria:

1. The patient is at least 18 years of age,
2. was initially diagnosed with peri-implantitis at ≥1 implant (peri-implant probing depth (PPD) ≥ 6 mm together with bleeding and/or suppuration on probing (BOP/SoP) and radiologically assessed marginal bone loss ≥ 3 mm),
3. had received treatment for peri-implantitis at least 5 years ago at the Graduate Clinic of Periodontics at University of Michigan, and
4. documentation from ≥ 5 years of clinical and radiological follow-up is available from U of M patients records.

Exclusion Criteria:

1. Has received or is currently receiving radiotherapy,
2. are currently pregnant, unsure of their pregnancy status, or are lactating (as reported by the patient),
3. has health condition(s) or takes medication(s) that are known to affect soft tissue or bone (e.g., Phenytoin)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects who were diagnosed with peri-implantitis and received treatment at least 5 years ago.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2018-12-04 (Actual); Primary Completion 2020-02-13 (Actual); Study Completion 2020-02-13 (Actual)

PRIMARY OUTCOMES:
Therapeutic resolution of the peri-implantitis as measured by radiographic bone loss | At least five years after the implant was treated for peri-implantitis
  The implant has no further radiographic bone loss when compared to previous radiographs.
Therapeutic resolution of the peri-implantitis as measured by erythema | At least five years after the implant was treated for peri-implantitis
  The implant has no current erythema of the peri-implant mucosa.
Therapeutic resolution of the peri-implantitis as measured by probing depths | At least five years after the implant was treated for peri-implantitis
  The implant has probing depths less than or equal to 5 millimeters.
Survival rate of the peri-implantitis treated dental implants | At least five years after the implant was treated for peri-implantitis
  Survival rate will be determined by the duration of implant survival (functioning, non-symptomatic implant after peri-implantitis treatment).

CONTACTS AND LOCATIONS:
Overall Officials: Hom-Lay Wang, DDS MSD PhD, Principal Investigator — Department of Periodontics and Oral Medicine University of Michigan
Locations (1):
- University of Michigan School of Dentistry, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Peri-implant mucositis and peri-implantitis: a current understanding of their diagnoses and clinical implications. J Periodontol. 2013 Apr;84(4):436-43. doi: 10.1902/jop.2013.134001. No abstract available. PMID 23537178
- [Background] Lindhe J, Meyle J; Group D of European Workshop on Periodontology. Peri-implant diseases: Consensus Report of the Sixth European Workshop on Periodontology. J Clin Periodontol. 2008 Sep;35(8 Suppl):282-5. doi: 10.1111/j.1600-051X.2008.01283.x. PMID 18724855
- [Background] Lang NP, Berglundh T; Working Group 4 of Seventh European Workshop on Periodontology. Periimplant diseases: where are we now?--Consensus of the Seventh European Workshop on Periodontology. J Clin Periodontol. 2011 Mar;38 Suppl 11:178-81. doi: 10.1111/j.1600-051X.2010.01674.x. PMID 21323713
- [Background] Sanz M, Chapple IL; Working Group 4 of the VIII European Workshop on Periodontology. Clinical research on peri-implant diseases: consensus report of Working Group 4. J Clin Periodontol. 2012 Feb;39 Suppl 12:202-6. doi: 10.1111/j.1600-051X.2011.01837.x. PMID 22533957
- [Background] Derks J, Tomasi C. Peri-implant health and disease. A systematic review of current epidemiology. J Clin Periodontol. 2015 Apr;42 Suppl 16:S158-71. doi: 10.1111/jcpe.12334. PMID 25495683
- [Background] Mombelli A, Muller N, Cionca N. The epidemiology of peri-implantitis. Clin Oral Implants Res. 2012 Oct;23 Suppl 6:67-76. doi: 10.1111/j.1600-0501.2012.02541.x. PMID 23062130
- [Background] Kotsovilis S, Karoussis IK, Trianti M, Fourmousis I. Therapy of peri-implantitis: a systematic review. J Clin Periodontol. 2008 Jul;35(7):621-9. doi: 10.1111/j.1600-051X.2008.01240.x. Epub 2008 May 11. PMID 18476998
- [Background] Klokkevold PR, Han TJ. How do smoking, diabetes, and periodontitis affect outcomes of implant treatment? Int J Oral Maxillofac Implants. 2007;22 Suppl:173-202. PMID 18437796
- [Background] Canullo L, Penarrocha M, Monje A, Catena A, Wang HL, Penarrocha D. Association Between Clinical and Microbiologic Cluster Profiles and Peri-implantitis. Int J Oral Maxillofac Implants. 2017 Sep/Oct;32(5):1054-1064. doi: 10.11607/jomi.6043. PMID 28906504
- [Background] Machtei EE. Treatment Alternatives to Negotiate Peri-Implantitis. Adv Med. 2014;2014:487903. doi: 10.1155/2014/487903. Epub 2014 Jun 15. PMID 26556414
- [Background] Renvert S, Polyzois I, Claffey N. Surgical therapy for the control of peri-implantitis. Clin Oral Implants Res. 2012 Oct;23 Suppl 6:84-94. doi: 10.1111/j.1600-0501.2012.02554.x. PMID 23062132
- [Background] Romeo E, Lops D, Chiapasco M, Ghisolfi M, Vogel G. Therapy of peri-implantitis with resective surgery. A 3-year clinical trial on rough screw-shaped oral implants. Part II: radiographic outcome. Clin Oral Implants Res. 2007 Apr;18(2):179-87. doi: 10.1111/j.1600-0501.2006.01318.x. PMID 17348882
- [Background] Wiltfang J, Zernial O, Behrens E, Schlegel A, Warnke PH, Becker ST. Regenerative treatment of peri-implantitis bone defects with a combination of autologous bone and a demineralized xenogenic bone graft: a series of 36 defects. Clin Implant Dent Relat Res. 2012 Jun;14(3):421-7. doi: 10.1111/j.1708-8208.2009.00264.x. Epub 2010 Feb 3. PMID 20132246
- [Background] Khoury F, Buchmann R. Surgical therapy of peri-implant disease: a 3-year follow-up study of cases treated with 3 different techniques of bone regeneration. J Periodontol. 2001 Nov;72(11):1498-508. doi: 10.1902/jop.2001.72.11.1498. PMID 11759861
- [Background] Li X, Wang X, Zhao T, Gao B, Miao Y, Zhang D, Dong Y. Guided bone regeneration using chitosan-collagen membranes in dog dehiscence-type defect model. J Oral Maxillofac Surg. 2014 Feb;72(2):304.e1-14. doi: 10.1016/j.joms.2013.09.042. Epub 2013 Oct 9. PMID 24438600
- [Background] Schou S, Holmstrup P, Skovgaard LT, Stoltze K, Hjorting-Hansen E, Gundersen HJ. Autogenous bone graft and ePTFE membrane in the treatment of peri-implantitis. II. Stereologic and histologic observations in cynomolgus monkeys. Clin Oral Implants Res. 2003 Aug;14(4):404-11. doi: 10.1034/j.1600-0501.2003.120910.x. PMID 12869002
- [Background] Schou S, Holmstrup P, Jorgensen T, Stoltze K, Hjorting-Hansen E, Wenzel A. Autogenous bone graft and ePTFE membrane in the treatment of peri-implantitis. I. Clinical and radiographic observations in cynomolgus monkeys. Clin Oral Implants Res. 2003 Aug;14(4):391-403. doi: 10.1034/j.1600-0501.2003.120909.x. PMID 12869001
- [Background] Javed F, Al-Askar M, Al-Rasheed A, Al-Hezaimi K. Significance of the platelet-derived growth factor in periodontal tissue regeneration. Arch Oral Biol. 2011 Dec;56(12):1476-84. doi: 10.1016/j.archoralbio.2011.06.020. Epub 2011 Jul 20. PMID 21774915
- [Background] Jung RE, Glauser R, Scharer P, Hammerle CH, Sailer HF, Weber FE. Effect of rhBMP-2 on guided bone regeneration in humans. Clin Oral Implants Res. 2003 Oct;14(5):556-68. doi: 10.1034/j.1600-0501.2003.00921.x. PMID 12969359
- [Background] Froum SJ, Rosen PS. A proposed classification for peri-implantitis. Int J Periodontics Restorative Dent. 2012 Oct;32(5):533-40. PMID 22754901
- [Background] Faggion CM Jr, Listl S, Tu YK. Assessment of endpoints in studies on peri-implantitis treatment--a systematic review. J Dent. 2010 Jun;38(6):443-50. doi: 10.1016/j.jdent.2010.03.003. Epub 2010 Mar 11. PMID 20226832
- [Background] Roos-Jansaker AM, Lindahl C, Persson GR, Renvert S. Long-term stability of surgical bone regenerative procedures of peri-implantitis lesions in a prospective case-control study over 3 years. J Clin Periodontol. 2011 Jun;38(6):590-7. doi: 10.1111/j.1600-051X.2011.01729.x. Epub 2011 Apr 13. PMID 21488935
- [Background] Berglundh T, Armitage G, Araujo MG, Avila-Ortiz G, Blanco J, Camargo PM, Chen S, Cochran D, Derks J, Figuero E, Hammerle CHF, Heitz-Mayfield LJA, Huynh-Ba G, Iacono V, Koo KT, Lambert F, McCauley L, Quirynen M, Renvert S, Salvi GE, Schwarz F, Tarnow D, Tomasi C, Wang HL, Zitzmann N. Peri-implant diseases and conditions: Consensus report of workgroup 4 of the 2017 World Workshop on the Classification of Periodontal and Peri-Implant Diseases and Conditions. J Periodontol. 2018 Jun;89 Suppl 1:S313-S318. doi: 10.1002/JPER.17-0739. PMID 29926955
- [Background] Schwarz F, Herten M, Sager M, Bieling K, Sculean A, Becker J. Comparison of naturally occurring and ligature-induced peri-implantitis bone defects in humans and dogs. Clin Oral Implants Res. 2007 Apr;18(2):161-70. doi: 10.1111/j.1600-0501.2006.01320.x. PMID 17348880
- [Background] Monje A, Wang HL, Nart J. Association of Preventive Maintenance Therapy Compliance and Peri-Implant Diseases: A Cross-Sectional Study. J Periodontol. 2017 Oct;88(10):1030-1041. doi: 10.1902/jop.2017.170135. Epub 2017 May 26. PMID 28548886